CLINICAL TRIAL: NCT05477732
Title: Effects of Bifidobacterium Longum OLP-01 Supplement on Cognitive Function, Exercise Performance, Nutritional Status and Gut Microbiota in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N202011038
Record Dates: First submitted 2022-07-18; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Stroke
Keywords: Bifidobacterium longum OLP-01; Stroke; Cognitive function; Exercise performance; Nutritional status; Gut microbiota
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): Subjects in placebo group will treat with placebo.
  Interventions: Other: Placebo
- Supplement group (Experimental): Subjects in supplement group will treat with Bifidobacterium longum OLP-01.
  Interventions: Dietary Supplement: Bifidobacterium longum OLP-01

INTERVENTIONS:
Dietary Supplement: Bifidobacterium longum OLP-01 — Bifidobacterium longum OLP-01 is one of probiotics. Subjects in OLP-01 group will supplement with either 2 × 1010 colony-forming unit (CFU) of Bifidobacterium longum OLP-01 powder per day for 12 weeks.
  Arms: Supplement group
Other: Placebo — Subjects in placebo group will supplement with placebo powder per day for 12 weeks.
  Arms: Placebo group

SUMMARY:
Stroke is a syndrome of acute, focal neurological deficit attributed to vascular injury of the central nervous system. It was the 2nd leading cause of death worldwide and accompanied by high disability rate also increases the social burden.Our research is to investigate the effects of intervention with Bifidobacterium longum OLP-01 on cognitive function, exercise performance, nutritional status and gut microbiota in stroke patients.

1. Study population:

   We will recruit 120 stroke patients and the inclusion criteria are: (1) Aged 20-75 years old, (2) Diagnosed with stroke more than 3 months, (3) Undergoing outpatient rehabilitation and the condition is stable. The exclusion criteria are: (1) Aphasia, dementia or depression, (2) BMI ≥ 35 kg/m2, (3) Cancer treatment in 3 months, (4) Some severe disease may interfere patients to join the study, (5) Failed to cooperate the examination and treatment because of emotion or mental condition.
2. Study design:

A two-arm single-blind randomized controlled clinical trial will be performed for 12 weeks and the subjects will be divided in to 2 groups: (1) placebo group, (2) supplement group. Subjects were asked to supplement with either 2 × 1010 colony-forming unit (CFU) of Bifidobacterium longum OLP-01 powder per day or placebo for 12 weeks. Medical history, drug use and life style questionnaires were giving before intervention. Outcomes will be assess in week 0 and week 12 during intervention.

3. Outcome assessment:

1. Anthropometry data: height, weight, body mass index, waist circumference, mid-upper arm circumference, hip circumference, calf circumference, waist to hip ratio.
2. Body composition: muscle mass, body fat, basal metabolic rate.
3. Clinical data: blood pressure, stroke related characteristics.
4. Blood biochemistry:

   A. Nutritional status: albumin, prealbumin, transferrin.

   B. Glycemic profiles: fasting blood glucose, glycated hemoglobin A1c (HbA1c).

   C. Lipid profiles: total cholesterol (TC), high density lipoprotein cholesterol (HDL-C), low density lipoprotein cholesterol (LDL-C), triglycerides (TG).

   D. Complete blood counts: white blood cells (WBC), red blood cells (RBC), hemoglobin (HB), platelet count (PLT), hematocrit (HCT), mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC).

   E. WBC differential counts: neutrophils (NEUT), lymphocytes (LYM), monocytes (MONO), eosinophils (EOS), basophils (BASO).

   F. C-reactive protein (CRP), interleukin-6 (IL-6), interleukin-10 (IL-10) and tumor necrosis factor alpha (TNF-α).
5. Gut microbiota: relative abundance, α-diversity, β-diversity.
6. Nutritional status: 3-day dietary record, mini-nutritional assessment (MNA).
7. Cognitive function: Montreal cognitive assessment (MoCA), trail-making test A and B (TMT A and B), Stroop color naming test.
8. Exercise performance: timed up and go test (TUGT), 6-min walking test.

The purpose of the study is to investigate the intervention of Bifidobacterium longum OLP-01 supplement on cognitive function, physiological performance, nutritional status, and gut microbiota in stroke patients.

ELIGIBILITY:
Inclusion criteria

* Aged 20-75 years old
* Diagnosed with stroke more than 3 months
* Undergoing outpatient rehabilitation and the condition is stable

Exclusion criteria

* Aphasia, dementia or depression
* BMI ≥ 35 kg/m2
* Cancer treatment in 3 months
* Some severe disease may interfere patients to join the study
* Failed to cooperate the examination and treatment because of emotion or mental condition.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-02-12 (Actual); Primary Completion 2023-02-11 (Estimated); Study Completion 2023-02-11 (Estimated)

PRIMARY OUTCOMES:
Montreal cognitive assessment (MoCA) | Week 0
  Cognitive function
Montreal cognitive assessment (MoCA) | Week 12
  Cognitive function
Montreal cognitive assessment (MoCA) (change) | Change from week 0 to week 12
  Cognitive function
Trail-making test A and B (TMT A and B) | Week 0
  Cognitive function
Trail-making test A and B (TMT A and B) | Week 12
  Cognitive function
Trail-making test A and B (TMT A and B) (change) | Change from week 0 to week 12
  Cognitive function
Stroop color naming test | Week 0
  Cognitive function
Stroop color naming test | Week 12
  Cognitive function
Stroop color naming test (change) | Change from week 0 to week 12
  Cognitive function
Timed up and go test (TUGT) | Week 0
  Exercise performance
Timed up and go test (TUGT) | Week 12
  Exercise performance
Timed up and go test (TUGT) (change) | Change from week 0 to week 12
  Exercise performance
6-min walking test | Week 0
  Exercise performance
6-min walking test | Week 12
  Exercise performance
6-min walking test (change) | Change from week 0 to week 12
  Exercise performance
Albumin | Week 0
  Nutritional Status
Albumin | Week 12
  Nutritional Status
Albumin (change) | Change from week 0 to week 12
  Nutritional Status
Pre-albumin | Week 0
  Nutritional Status
Pre-albumin | Week 12
  Nutritional Status
Pre-albumin (change) | Change from week 0 to week 12
  Nutritional Status
Transferrin | Week 0
  Nutritional Status
Transferrin | Week 12
  Nutritional Status
Transferrin (change) | Change from week 0 to week 12
  Nutritional Status
3-day dietary record | Week 0
  Nutritional Status
3-day dietary record | Week 12
  Nutritional Status
3-day dietary record (change) | Change from week 0 to week 12
  Nutritional Status
Mini-nutritional assessment (MNA) | Week 0
  Nutritional Status
Mini-nutritional assessment (MNA) | Week 12
  Nutritional Status
Mini-nutritional assessment (MNA) (change) | Change from week 0 to week 12
  Nutritional Status
Relative abundance | Week 0
  Gut microbiota Use the 16s RNA sequencing to conduct the next generation sequencing (NGS) measure the relative abundance, including the phylum, class, family, genus.
Relative abundance | Week 12
  Gut microbiota Use the 16s RNA sequencing to conduct the next generation sequencing (NGS) measure the relative abundance, including the phylum, class, family, genus.
α-diversity | Week 0
  Gut microbiota
α-diversity | Week 12
  Gut microbiota
β-diversity | Week 0
  Gut microbiota
β-diversity | Week 12
  Gut microbiota

SECONDARY OUTCOMES:
Height | Week 0
  Anthropometry data
Height | Week 12
  Anthropometry data
Height (change) | Change from week 0 to week 12
  Anthropometry data
Weight | Week 0
  Anthropometry data
Weight | Week 12
  Anthropometry data
Weight (change) | Change from week 0 to week 12
  Anthropometry data
Body mass index (BMI) | Week 0
  Anthropometry data Weight and height will be combined to report BMI in kg/m^2
Body mass index (BMI) | Week 12
  Anthropometry data Weight and height will be combined to report BMI in kg/m^2
Body mass index (BMI) (change) | Change from week 0 to week 12
  Anthropometry data Weight and height will be combined to report BMI in kg/m^2
Waist circumference | Week 0
  Anthropometry data
Waist circumference | Week 12
  Anthropometry data
Waist circumference (change) | Change from week 0 to week 12
  Anthropometry data
Mid-upper arm circumference | Week 0
  Anthropometry data
Mid-upper arm circumference | Week 12
  Anthropometry data
Mid-upper arm circumference (change) | Change from week 0 to week 12
  Anthropometry data
Hip circumference | Week 0
  Anthropometry data
Hip circumference | Week 12
  Anthropometry data
Hip circumference (change) | Change from week 0 to week 12
  Anthropometry data
Calf circumference | Week 0
  Anthropometry data
Calf circumference | Week 12
  Anthropometry data
Calf circumference (change) | Change from week 0 to week 12
  Anthropometry data
Waist to hip ratio | Week 0
  Anthropometry data Waist circumference and hip circumference will be combined to report waist to hip ratio
Waist to hip ratio | Week 12
  Anthropometry data Waist circumference and hip circumference will be combined to report waist to hip ratio
Waist to hip ratio (change) | Change from week 0 to week 12
  Anthropometry data Waist circumference and hip circumference will be combined to report waist to hip ratio
Muscle mass | Week 0
  Body composition
Muscle mass | Week 12
  Body composition
Muscle mass (change) | Change from week 0 to week 12
  Body composition
Body fat | Week 0
  Body composition
Body fat | Week 12
  Body composition
Body fat (change) | Change from week 0 to week 12
  Body composition
Basal metabolic rate | Week 0
  Body composition
Basal metabolic rate | Week 12
  Body composition
Basal metabolic rate (change) | Change from week 0 to week 12
  Body composition
Blood pressure | Week 0
  Clinical data
Blood pressure | Week 12
  Clinical data
Blood pressure (change) | Change from week 0 to week 12
  Clinical data
Stroke related characteristics (including the time since stroke diagnosed, side of lesion, stroke type, use of aid) | Week 0
  Stroke related characteristics would collect form clinical data or ask form subjects directly
Stroke related characteristics (including the time since stroke diagnosed, side of lesion, stroke type, use of aid) | Week 12
  Stroke related characteristics would collect form clinical data or ask form subjects directly
Medical history, drug use and life style questionnaires | Week 0
  Clinical data This questionnaires including 3 parts (medical history, drug use and life style). Medical history and drug use will write by subjects. Life style (e.g. smocking habit, exercise frequency) will ask the subjects.
Medical history, drug use and life style questionnaires | Week 12
  Clinical data This questionnaires including 3 parts (medical history, drug use and life style). Medical history and drug use will write by subjects. Life style (e.g. smocking habit, exercise frequency) will ask the subjects.
Fasting blood glucose | Week 0
  Blood biochemistry
Fasting blood glucose | Week 12
  Blood biochemistry
Fasting blood glucose (change) | Change from week 0 to week 12
  Blood biochemistry
Glycated hemoglobin A1c (HbA1c) | Week 0
  Blood biochemistry
Glycated hemoglobin A1c (HbA1c) | Week 12
  Blood biochemistry
Glycated hemoglobin A1c (HbA1c) (change) | Change from week 0 to week 12
  Blood biochemistry
Total cholesterol (TC) | Week 0
  Blood biochemistry
Total cholesterol (TC) | Week 12
  Blood biochemistry
Total cholesterol (TC) (change) | Change from week 0 to week 12
  Blood biochemistry
High density lipoprotein cholesterol (HDL-C) | Week 0
  Blood biochemistry
High density lipoprotein cholesterol (HDL-C) | Week 12
  Blood biochemistry
High density lipoprotein cholesterol (HDL-C) (change) | Change from week 0 to week 12
  Blood biochemistry
Low density lipoprotein cholesterol (LDL-C) | Week 0
  Blood biochemistry
Low density lipoprotein cholesterol (LDL-C) | Week 12
  Blood biochemistry
Low density lipoprotein cholesterol (LDL-C) (change) | Change from week 0 to week 12
  Blood biochemistry
Triglycerides (TG) | Week 0
  Blood biochemistry
Triglycerides (TG) | Week 12
  Blood biochemistry
Triglycerides (TG) (change) | Change from week 0 to week 12
  Blood biochemistry
White blood cells (WBC) | Week 0
  Blood biochemistry
White blood cells (WBC) | Week 12
  Blood biochemistry
White blood cells (WBC) (change) | Change from week 0 to week 12
  Blood biochemistry
Red blood cells (RBC) | Week 0
  Blood biochemistry
Red blood cells (RBC) | Week 12
  Blood biochemistry
Red blood cells (RBC) (change) | Change from week 0 to week 12
  Blood biochemistry
Hemoglobin (HB) | Week 0
  Blood biochemistry
Hemoglobin (HB) | Week 12
  Blood biochemistry
Hemoglobin (HB) (change) | Change from week 0 to week 12
  Blood biochemistry
Platelet count (PLT) | Week 0
  Blood biochemistry
Platelet count (PLT) | Week 12
  Blood biochemistry
Platelet count (PLT) (change) | Change from week 0 to week 12
  Blood biochemistry
Hematocrit (HCT) | Week 0
  Blood biochemistry
Hematocrit (HCT) | Week 12
  Blood biochemistry
Hematocrit (HCT) (change) | Change from week 0 to week 12
  Blood biochemistry
Mean corpuscular volume (MCV) | Week 0
  Blood biochemistry
Mean corpuscular volume (MCV) | Week 12
  Blood biochemistry
Mean corpuscular volume (MCV) (change) | Change from week 0 to week 12
  Blood biochemistry
Mean corpuscular hemoglobin (MCH) | Week 0
  Blood biochemistry
Mean corpuscular hemoglobin (MCH) | Week 12
  Blood biochemistry
Mean corpuscular hemoglobin (MCH) (change) | Change from week 0 to week 12
  Blood biochemistry
Mean corpuscular hemoglobin concentration (MCHC) | Week 0
  Blood biochemistry
Mean corpuscular hemoglobin concentration (MCHC) | Week 12
  Blood biochemistry
Mean corpuscular hemoglobin concentration (MCHC) (change) | Change from week 0 to week 12
  Blood biochemistry
Neutrophils (NEUT) | Week 0
  Blood biochemistry (WBC counts)
Neutrophils (NEUT) | Week 12
  Blood biochemistry (WBC counts)
Neutrophils (NEUT) | Change from week 0 to week 12
  Blood biochemistry (WBC counts)
Lymphocytes (LYM) | Week 0
  Blood biochemistry (WBC counts)
Lymphocytes (LYM) | Week 12
  Blood biochemistry (WBC counts)
Lymphocytes (LYM) | Change from week 0 to week 12
  Blood biochemistry (WBC counts)
Monocytes (MONO) | Week 0
  Blood biochemistry (WBC counts)
Monocytes (MONO) | Week 12
  Blood biochemistry (WBC counts)
Monocytes (MONO) | Change from week 0 to week 12
  Blood biochemistry (WBC counts)
Eosinophils (EOS) | Week 0
  Blood biochemistry (WBC counts)
Eosinophils (EOS) | Week 12
  Blood biochemistry (WBC counts)
Eosinophils (EOS) | Change from week 0 to week 12
  Blood biochemistry (WBC counts)
Basophils (BASO) | Week 0
  Blood biochemistry (WBC counts)
Basophils (BASO) | Week 12
  Blood biochemistry (WBC counts)
Basophils (BASO) | Change from week 0 to week 12
  Blood biochemistry (WBC counts)
Interleukin-6 (IL-6), interleukin-10 (IL-10), tumor necrosis factor alpha (TNF-α) | Week 0
  Blood biochemistry (cytokines)
Interleukin-6 (IL-6), interleukin-10 (IL-10), tumor necrosis factor alpha (TNF-α) | Week 12
  Blood biochemistry (cytokines)
Interleukin-6 (IL-6), interleukin-10 (IL-10), tumor necrosis factor alpha (TNF-α) (change) | Change from week 0 to week 12
  Blood biochemistry (cytokines)
C-reactive protein (CRP) | Week 0
  Blood biochemistry
C-reactive protein (CRP) | Week 12
  Blood biochemistry
C-reactive protein (CRP) (change) | Change from week 0 to week 12
  Blood biochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Chao Jane C-J, PhD, Principal Investigator — Taipei Medical University, Taiwan, R.O.C.
Locations (3):
- Taiwan (3):
  - Department of rehabilitation, ShuangHo Hospital, New Taipei City
  - Department of rehabilitation, Taipei Medical University Hospital, Taipei
  - Department of rehabilitation, WanFang Hospital, Taipei